CLINICAL TRIAL: NCT06532279
Title: A Randomized, Masked, Placebo Controlled, Phase II Trial Of Concurrent Chemoradiation With BMX-001 In Patients With Head And Neck Squamous Cell Carcinoma Receiving Concurrent Chemoradiation
Brief Title: Testing the Addition of the Drug BMX-001, a Radioprotector, or a Placebo to the Usual Chemoradiation Therapy for Patients With Head and Neck Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NRG-CC013; NCI-2024-03906 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-CC013 (Other: NRG Oncology); NRG-CC013 (Other: DCP); NRG-CC013 (Other: CTEP); UG1CA189867 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Head and Neck Squamous Cell Carcinoma; Hypopharyngeal Squamous Cell Carcinoma; Laryngeal Squamous Cell Carcinoma; Nasopharyngeal Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Oropharyngeal Squamous Cell Carcinoma; Stage 0 Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage 0 Hypopharyngeal Carcinoma AJCC v8; Stage 0 Nasopharyngeal Carcinoma AJCC v8; Stage 0 Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage I Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage I Hypopharyngeal Carcinoma AJCC v8; Stage I Laryngeal Cancer AJCC v8; Stage I Lip and Oral Cavity Cancer AJCC v8; Stage I Nasopharyngeal Carcinoma AJCC v8; Stage I Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage II Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage II Hypopharyngeal Carcinoma AJCC v8; Stage II Laryngeal Cancer AJCC v8; Stage II Lip and Oral Cavity Cancer AJCC v8; Stage II Nasopharyngeal Carcinoma AJCC v8; Stage II Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage III Head and Neck Cutaneous Squamous Cell Carcinoma AJCC v8; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Nasopharyngeal Carcinoma AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVA Hypopharyngeal Carcinoma AJCC v8; Stage IVA Laryngeal Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8; Stage IVA Nasopharyngeal Carcinoma AJCC v8; Stage IVA Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IVB Hypopharyngeal Carcinoma AJCC v8; Stage IVB Laryngeal Cancer AJCC v8; Stage IVB Lip and Oral Cavity Cancer AJCC v8; Stage IVB Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stomatitis
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Nasopharyngeal Carcinoma; Carcinoma; Laryngeal Neoplasms; Mouth Neoplasms; Stomatitis | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Mn(III) meso-tetrakis(N-n-butoxyethylpyridinium-2-yl)porphyrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind. Fully blinded team members- Refers to individuals that have no access to view preparation of study drug. Study team members who are administering study drug (not preparing) will be included, however individuals that administer study drug should not perform efficacy assessments.
  Any investigator or sub-investigator involved in performing efficacy and safety assessments- These individuals should not be involved in preparation of the study drug and should avoid visual access during study drug administration when possible. Where possible, any other site staff member who does not have specific responsibilities that require access to IP (e.g., data entry assistant) should remain fully blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (placebo) (Placebo Comparator): Patients receive cisplatin QW or Q3W and undergo image-guided intensity-modulated radiation therapy QD 5 days per week for 7 weeks per SOC. In addition to usual symptom management, patients receive placebo SC as early as 96 hours and no later than one hour prior to their first dose of radiation therapy, and as early as 96 hours and no later than 48 hours prior to first dose of cisplatin. Patients then receive placebo SC BIW for 8 weeks (16 doses). Patients also undergo CT and/or MRI on study and may optionally undergo collection of blood, serum, and/or plasma throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: Placebo Administration; Other: Questionnaire Administration
- Arm 2 (BMX-001) (Experimental): Patients receive cisplatin QW or Q3W and undergo image-guided intensity-modulated radiation therapy QD 5 days per week for 7 weeks per SOC. In addition to usual symptom management, patients receive BMX-001 SC as early as 96 hours and no later than one hour prior to their first dose of radiation therapy, and as early as 96 hours and no later than 48 hours prior to first dose of cisplatin. Patients then receive BMX-001 SC BIW for 8 weeks (16 doses). Patients also undergo CT and/or MRI on study and may optionally undergo collection of blood, serum, and/or plasma throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: MnSOD Mimetic BMX-001; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual symptom management
  Other Names: standard of care; standard therapy
Procedure: Biospecimen Collection — Undergo collection of blood, serum, and/or plasma samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given cisplatin
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Image Guided Radiation Therapy — Undergo image-guided radiation therapy
  Other Names: IGRT; Image Guided Radiotherapy; image-guided radiation therapy; Image-Guided Radiotherapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo intensity-modulated radiation therapy
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: MnSOD Mimetic BMX-001 — Given SC
  Other Names: BMX-001; Manganese (III) ortho N-Butoxyethylpyridylporphyrin; Manganese Butoxyethyl Pyridyl Porphyrin; Mitochondrial Manganese Superoxide Dismutatse Mimetic BMX-001; Mn(III) meso-tetrakis(N-n-butoxyethylpyridinium-2-yl)porphyrin; MnTnBuOE-3-PyP 5+
  Arms: Arm 2 (BMX-001)
Drug: Placebo Administration — Given SC
  Arms: Arm 1 (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial compares the effectiveness of adding BMX-001 to usual symptom management versus usual symptom management alone for reducing oral mucositis in patients who are receiving chemoradiation for head and neck cancer. Oral mucositis (inflammation and mouth sores) is a common side effect of chemoradiation that can cause pain and difficulty swallowing. Usual management of these side effects typically consists of using mouth rinses and pain medications during treatment and for several weeks after completion of treatment. BMX-001 neutralizes harmful substances in the body, preventing damage to macromolecules such as DNA and minimizes free radical-related toxicity in normal tissues. Adding BMX-001 to usual symptom management may be more effective than usual symptom management alone at reducing oral mucositis in patients receiving chemoradiation for head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the incidence of severe oral mucositis (SOM) between manganese superoxide dismutase (MnSOD) mimetic BMX-001 (BMX-001) and placebo, defined as >= grade 3 per World Health Organization (WHO) criteria from the start of radiation through 4 weeks after completion of study treatment, with additional assessments at 6, 8 and 12 weeks after completion of study treatment.

SECONDARY OBJECTIVES:

I. To compare the duration of SOM in the BMX-001 arm versus (vs.) placebo arm. II. To assess the difference between arms in the Oral Mucositis Weekly Questionnaire-Head and Neck (OMWQ-HN) change score from baseline to 4 weeks after the end of chemoradiation.

III. To describe the incidence and severity of xerostomia and radiation dermatitis, as measured by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0, in both arms.

IV. To compare the duration of radiation dermatitis in the BMX-001 arm vs. placebo arm.

V. To describe toxicity, as measured by CTCAE v5.0 and Patient Reported Outcome (PRO)-CTCAE, in both arms.

EXPLORATORY OBJECTIVES:

I. To assess the between arm difference in progression-free survival (PFS). II. To assess the between arm difference in overall survival (OS). III. Data demonstrating improvement in pain, as measured by reduction in narcotic use between BMX-001 versus usual care.

IV. Collect serum and plasma for future translational research analyses.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive cisplatin once weekly (QW) or once every 3 weeks (Q3W) and undergo image-guided intensity-modulated radiation therapy once daily (QD) 5 days per week for 7 weeks per standard of care (SOC). In addition to usual symptom management, patients receive placebo subcutaneously (SC) as early as 96 hours and no later than one hour prior to their first dose of radiation therapy, and as early as 96 hours and no later than 48 hours prior to first dose of cisplatin. Patients then receive placebo SC twice a week (BIW) for 8 weeks (16 doses). Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) on study and may optionally undergo collection of blood, serum, and/or plasma throughout the study.

ARM 2: Patients receive cisplatin QW or Q3W and undergo image-guided intensity-modulated radiation therapy QD 5 days per week for 7 weeks per SOC. In addition to usual symptom management, patients receive BMX-001 SC as early as 96 hours and no later than one hour prior to their first dose of radiation therapy, and as early as 96 hours and no later than 48 hours prior to first dose of cisplatin. Patients then receive BMX-001 SC BIW for 8 weeks (16 doses). Patients also undergo CT and/or MRI on study and may optionally undergo collection of blood, serum, and/or plasma throughout the study.

After completion of study treatment, patients are followed up at 1, 2, 3, 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be planned to receive radiation and concurrent cisplatin chemotherapy as definitive therapy. Patients planned to receive concurrent cisplatin and radiation therapy in the adjuvant setting are not eligible.
* At least two subsites (buccal mucosa, lips, retromolar trigone, floor of mouth, oral tongue, tonsil, soft palate, or hard palate) must have at least 1cc or 1% of the subsite volume receiving >= 50 Gy. In cases of uncertainty, the enrolling clinician can ensure coverage by inspecting the 50 Gy isodose line and using the table describing the anatomic boundaries of the individual subsites contained within the extended cavity contour. The two or more subsites receiving >= 50 Gy must be documented by the enrolling physician.
* Pathologically confirmed (histologically or cytologically) squamous cell carcinoma of the oropharynx, larynx, hypopharynx, nasopharynx, or oral cavity.
* P16 and/or human papillomavirus (HPV) status (via polymerase chain reaction [PCR] or in situ hybridization [ISH]) must be documented for patients with oropharynx cancer.
* No patients with T0/Tx/unknown primary disease.
* No definitive clinical or radiologic evidence of metastatic (M1) disease related to current diagnosis.
* Able to receive intensity-modulated radiation therapy (IMRT) delivered as daily fractions of 2.0 Gy once per weekday with a cumulative radiation dose of 70 Gy.
* Age >= 18.
* Zubrod performance status of 0-2.
* Potassium ≥ institutional lower limit of normal (LLN) and magnesium ≥ institutional LLN. Oral or intravenous (IV) replacement therapy of potassium or magnesium is permitted if parameters can be met after repletion.
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3.
* Platelets >= 100,000 cells/mm^3.
* Hemoglobin >= 9.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 10.0 g/dl is acceptable).
* Adequate renal function defined as creatinine clearance (CrCL) > 50 mL/min by the Cockcroft-Gault formula.
* Total bilirubin =< 2 x institutional upper limit of normal (ULN) (not applicable to patients with known Gilbert's syndrome).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN.
* No prior radiotherapy that would result in overlap of radiation treatment fields with planned treatment for study cancer, e.g., breast cancer with irradiation of the supraclavicular fossa/level 4 neck.
* No concurrent treatment with nitrates or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure.
* No prior history of gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease. In other words, to participate in this protocol, the patient must have clinically or radiographically evident gross disease for which disease response can be assessed.
* No current treatment of adjuvant post-operative (op) chemoradiation.
* No systemic treatment with inducers or strong inhibitors of cytochrome P450 =< 4 days before registration. Note: Patients undergoing steroid treatment as a component of the anti-emetic regimen for cisplatin are eligible for the study. Treatment with the antifungal medications, nystatin, fluconazole , miconazole and clotrimazole are allowed.
* No prior induction chemotherapy treatment.
* No prior unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ, basal cell skin carcinoma, resected T1-2N0M0 differentiated thyroid cancers, Ta bladder cancers, or low risk prostate cancer.
* No clinically significant hearing impairment that precludes cisplatin, as per physician assessment.
* No serious cardiovascular disease or cerebrovascular disease in the last 6 months prior to study enrollment; defined as a cerebrovascular accident, myocardial infarction, unstable angina, serious cardiac arrhythmia uncontrolled by medication or with the potential to interfere with protocol treatment, or current New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), or admission within last 6 months for CHF exacerbation; (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification).
* No valvular heart disease.
* No significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to enrollment.
* No history or evidence upon physical/neurological examination of central nervous system disease (e.g., seizures) unrelated to cancer unless adequately controlled by medication.
* No acute bacterial, viral, or fungal infection requiring intravenous antimicrobials within 7 days of enrollment.
* No history of chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration.
* No known personal or family history of long QT Syndrome; no marked baseline prolongation of QT/corrected QT (QTc) interval (i.e., ≥ 2 electrocardiograms [EKGs] in prior 3 months of a QTc interval > 450 milliseconds (ms) for males and > 470 ms for females using the specific/usual choice by clinical center for correction factor.
* Persistent grade 3-4 (CTCAE version 5.0) electrolyte abnormalities must be reversible to ≤ grade 1 with supplementation.
* No poorly controlled hypertension (systolic blood pressure [SBP] > 160 and/or diastolic blood pressure [DBP] > 95) over 2 repeated measures within 30 days prior to registration.
* No grade >= 2 oral mucositis per CTCAE version 5.0.
* No grade >= 2 hypotension per CTCAE v. 5.0.
* No medical necessity for anti-arrhythmics with significant risk of QTc prolongation such as class I and class III anti-arrhythmics. These include but are not limited to amiodarone, quinidine, dofetilide, sotalol, flecainide, and lidocaine.
* No medical necessity for medications listed as prohibited.

  * For standard management of oral mucositis, clinicians may consult the Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO) Clinical Practice Guidelines for the Management of Mucositis Secondary to Cancer Therapy. The only intervention against mucositis that is supported by level I evidence is low-level laser therapy (LLLT). Honey is rated at level II and benzydamine, which isn't available in the United States (US), is rated at level III. There are no other positively rated interventions.
  * LLLT is prohibited in this study as its availability remains limited, it is not Food and Drug Administration (FDA) approved in the US, and it is considered investigational in many circumstances requiring enrollment in a dedicated protocol who requirements could conflict with this one. Therefore, institutions that use LLLT should only enroll patients who would not be eligible for (or do not want) that intervention. Honey is not on the list of prohibited medications for this study. Given the MASCC recommendation, benzydamine is allowed, although there is lack of availability in the United States of America (USA). The other listed prohibited medications are not recommended by MASCC and some are potentially harmful, such as glutamine, which is associated with mortality in patients receiving stem cell transplant.
* No history of allergic reaction to the study agent(s), compounds of similar chemical or biologic composition to the study agent (s) (or any of its excipients).
* Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe oral mucositis (SOM) | From start of radiation through 4 weeks after completion of study treatment
  Proportion of patients with reported SOM >= grade 3 per World Health Organization criteria.

SECONDARY OUTCOMES:
Duration of SOM | Up to 12 weeks after completion of chemoradiation
  Defined from first determination of >= grade 3 oral mucositis (OM) to the first instance of non-SOM (=< grade 2), without subsequent instance of >= grade 3 within the following 4 weeks.
Time to SOM | Up to 12 weeks after completion of chemoradiation
  Defined from date of randomization to date of first determination of >= grade 3 OM.
Incidence and duration of xerostomia and radiation dermatitis | Up to 12 weeks after completion of chemoradiation
  The proportion of patients with any grade and grade ≥ 3 xerostomia and radiation dermatitis, separately. Duration is measured from the first determination of radiation dermatitis or xerostomia, separately, (grade ≥ 1 as measured by Common Terminology Criteria for Adverse Events [CTCAE] version [v] 5.0) to the first report of none (grade 0).
Incidence of toxicity | Up to 24 months after completion of chemoradiation
  Adverse events (AEs) will be graded by the physician-reported CTCAE v5.0 and also measured using the Patient Reported Outcome-CTCAE. Counts of all AEs by grade will be provided by treatment arm.
Patient reported oral mucositis | Up to 24 months after completion of chemoradiation
  Will be measured by the Oral Mucositis Weekly Questionnaire (OMWQ). Decline within patients is defined using a minimally important difference of 7.

OTHER OUTCOMES:
Pain improvement | Up to 24 months after completion of chemoradiation
  Pain improvement will be measured by opioid use collected in morphine equivalent doses.
Progression-free survival (PFS) | Up to 24 months after completion of chemoradiation
  PFS will be calculated from the date of randomization until occurrence of local, regional (neck lymph nodes) or distant failure, or death. PFS rates will be estimated using the Kaplan-Meier method. Patients without an event will be censored at their last disease assessment.
Overall survival (OS) | Up to 24 months after completion of chemoradiation
  OS will be calculated from the date of randomization to death and estimated using the Kaplan-Meier method. Patients alive without an event will be censored at their last known follow-up time.

CONTACTS AND LOCATIONS:
Overall Officials: David M Brizel, Principal Investigator — NRG Oncology
Locations (143):
- United States (143):
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Phoenix, Phoenix, Arizona
  - Arizona Center for Cancer Care - Scottsdale, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - Arizona Center for Cancer Care, Tempe, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Keck Medicine of USC Buena Park, Buena Park, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Shaw Cancer Center, Edwards, Colorado
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Sarasota Memorial Hospital-Venice, N. Venice, Florida
  - Moffitt Cancer Center at SouthShore, Ruskin, Florida
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Sarasota Memorial Health Care Center at University Parkway, Sarasota, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists - Venice Pinebrook, Venice, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Baptist Health Hardin, Elizabethtown, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Lancaster Radiation Therapy Center, Lancaster, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin